CLINICAL TRIAL: NCT02470520
Title: Observational Study Measuring Essential Nutrients in Critically Ill Patients With Severe Acute Kidney Injury Treated With and Without Continuous Haemofiltration
Brief Title: Essential Nutrients in Critically Ill Patients With Severe AKI Treated With and Without CRRT
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RJ113/N062
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Acute Kidney Failure
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AKI without CRRT: Patients with AKI who are not treated with continuous renal replacement therapy
- AKI with CRRT: Patients with AKI who are treated with continuous renal replacement therapy
  Interventions: Procedure: CRRT

INTERVENTIONS:
Procedure: CRRT — continuous renal replacement therapy
  Groups: AKI with CRRT

SUMMARY:
The aim of this study is to measure plasma levels of essential vitamins, trace elements and amino acids in critically ill patients with severe AKI. In patients who are treated with continuous renal replacement therapy, we plan to evaluate whether there are any additional losses of nutrients into the filtrate.

DETAILED DESCRIPTION:
Background: Critically ill patients with acute kidney injury (AKI) have a high risk of dying, especially if renal replacement therapy (RRT) is needed. It remains uncertain whether essential trace elements, vitamins and amino acids are lost during RRT in sufficient amounts to result in clinically significant deficiencies. At present, nutrition guidelines for patients with AKI on RRT do not account for any potential losses of micronutrients across the filter.

Hypothesis:

Critically ill patients with AKI have inadequate plasma nutrient levels. If continuous renal replacement therapy (CRRT) is required, there are additional losses of essential nutrients.

Aims:

To serially measure plasma levels of essential vitamins, trace elements and amino acids in critically ill patients with severe AKI and to evaluate whether there are any additional losses into the filtrate during CRRT

Objectives:

To perform serial measurements of plasma levels of selenium, zinc, copper, iron, vitamins B1, B6, B12, C and D, folic acid and essential amino acids in all patients with severe AKI and to measure any losses of the same nutrients in the filtrate in a cohort of patients on CRRT for >24 hours.

Patient population:

level 3 critically ill adult patients with severe AKI

Study size:

40 patients of whom 20 patients are treated with CRRT for >24 hours.

Study design:

observational non-interventional study in at least 2 large tertiary care centres in the United Kingdom

Outcomes:

Primary outcome: difference in plasma concentrations of essential trace elements and vitamins between patients with and without CRRT.

Secondary outcomes: a) concentrations of trace elements, vitamins and amino acids in filtrate in patients on CRRT; b) differences in filtrate losses between patients on CRRT ≤30ml/kg/hr versus >30ml/kg/hr.

Laboratory measurements:

Measurement of baseline plasma Selenium, Zinc, Copper, iron, Vitamins B1, B6, B12, C and D, folic acid and essential amino acids levels and repeat serial measurement of the same panel of nutrients in all patients for up to 6 days with additional concomitant measurement of nutrient levels in filtrate in cohort of patients on CRRT. In addition, daily measurement of serum electrolytes, liver profile, serum albumin and c-reactive protein.

Data collection:

Recording of the following potential confounders: type of nutrition, dose of CRRT, type of membrane.

Statistics:

Determination of the change in plasma nutrient levels over 6 days, and between baseline and 24 - 144 hours after initiation of CRRT. The estimates will be used to inform the design of an intervention study exploring the value of nutrient supplementation.

ELIGIBILITY:
Inclusion Criteria:

* adult patients in the Critical Care Unit with severe AKI

Exclusion Criteria:

* pre-existing dialysis dependent renal failure
* life expectancy <48 hours
* need for total parenteral nutrition
* need for supplementation with intravenous multivitamins or trace elements
* Jehovah's witness
* patients with haemoglobin <7g/dL (unless being transfused for clinical reasons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with severe acute kidney injury
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
serum levels of essential nutrients | up to 6 days

SECONDARY OUTCOMES:
levels of essential nutrients in filtrate | up to 6 days
  concentrations of trace elements, vitamins and amino acids in filtrate in patients on CRRT